CLINICAL TRIAL: NCT01467531
Title: A Phase 1, Open-Label, Crossover Study to Evaluate the Pharmacokinetics and Safety of GSK1265744 and Rilpivirine and Dolutegravir and Rilpivirine in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of GSK1265744 and Rilpivirine and Dolutegravir and Rilpivirine in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 116181
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Infections, Human Immunodeficiency Virus and Hepatitis
Keywords: HIV, GSK1265744, GSK1349572, dolutegravir, rilpivirine, drug interaction, pharmacokinetics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; Hepatitis | interventions — dolutegravir; Rilpivirine; cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Period 1 Treatment A = Dolutegravir 50mg q24h x 5 days; Period 2 Treatment B = Rilpivirine 25mg q24h x 11; Period 3 Dolutegravir 50mg q24h + Rilpivirine q24h x 5 days
  Interventions: Drug: Dolutegravir; Drug: Rlipivirine
- Cohort 2 (Experimental): Period 1 Treatment A = GSK1265744 30mg q24h x 12 days; Period 2 Treatment B = Rilpivirine 25mg q24h x 12; Period 3 GSK1265744 30mg q24h + Rilpivirine q24h x 12 days
  Interventions: Drug: Rlipivirine; Drug: GSK1265744

INTERVENTIONS:
Drug: Dolutegravir — 50mg q 24h
  Other Names: GSK1349572
  Arms: Cohort 1
Drug: Rlipivirine — 25mg q24h
  Other Names: Edurant
Drug: GSK1265744 — 30mg q24h
  Arms: Cohort 2

SUMMARY:
This will be a single-center, two-cohort, three-period study in healthy adult subjects. Approximately 16 healthy subjects will be enrolled in Cohort 1 to provide data from 14 evaluable subjects. Approximately 12 healthy subjects will be enrolled in Cohort 2 to provide data from 10 evaluable subjects. Subjects will have a screening visit within 30 days prior to the first dose of study drug, three treatment periods, and a follow-up visit 7-14 days after the last dose of study drug. There will be a washout period between Period 1 and Period 2 but no washout between Period 2 and Period 3. Day 1 of Period 3 will start the day after the last day in Period 2. The study will be conducted on an out-patient basis except for days where serial pharmacokinetic sampling and safety assessments are scheduled.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator feels that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol.
* Body weight greater than or equal to 50 kg for males and 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study as defined in the protocol.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetic Parameters following Dolutegravir administration with and without rilpivirine | Cohort 1: Period 1 and 3 on Day 5: pre-dose, 1, 2, 3, 4, 8, 12 and 24 hours post dose.
  Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC(0-tau)), Maximum observed concentration (Cmax), Time of occurrence of Cmax (tmax), Pre-dose (trough) concentration at the end of the dosing interval (Ctau)
Composite of Pharmacokinetic Parameters following GSK1265744 administration with and without rilpivirine | Cohort 2: Period 2 and 3, Day 12: pre-dose, 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24hrs post dose.
  steady state, AUC(0-t), Cmax, tmax, and Ctau
Composite of Pharmacokinetic Parameters following rilpivirine administration with and without Dolutegravir | Cohort 1: Period 2, Day 11: pre-dose, 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24hrs post dose. Period 3: Day 5 pre-dose 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24hrs post dose
  steady state, AUC(0-tau), Cmax, tmax, and Ctau
Composite of Pharmacokinetic Parameters following rilpivirine administration with and without GSK1265744 | Cohort 2: Periods 1 and 3: Day 12: pre-dose, 1, 2, 3, 4, 8, 12 and 24hrs post dose
  AUC(0-tau), Cmax, tmax, and Ctau

SECONDARY OUTCOMES:
Safety and tolerability parameters, including the collection of all adverse events | 42 days or final visit has occurred
  Collected from first dose to final visit.
Safety and tolerability parameters, including the collection of any concurrent medication from first dose to final visit | 42 days or final visit has occurred
  Collected from first dose to final visit.
Safety and tolerability parameters, including change from baseline in clinical laboratory tests (hematology, chemistry, urinalysis) assessments | 42 days or final assessment has occurred
Safety and tolerability parameters, including change from baseline in ECG assessments | 42 days or final assessment has occurred
Safety and tolerability parameters, including change from baseline in vital signs assessments | 42 days or final assessment has occurred

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Derived] Ford SL, Gould E, Chen S, Margolis D, Spreen W, Crauwels H, Piscitelli S. Lack of pharmacokinetic interaction between rilpivirine and integrase inhibitors dolutegravir and GSK1265744. Antimicrob Agents Chemother. 2013 Nov;57(11):5472-7. doi: 10.1128/AAC.01235-13. Epub 2013 Aug 26. PMID 23979733